CLINICAL TRIAL: NCT03074877
Title: Substance Use Screening and Prevention for Adolescents in Pediatric Primary Care
Acronym: SKY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01DA036628-02 (NIH)
Record Dates: First submitted 2017-02-13; First posted 2017-03-09 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Substance Use
Keywords: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Family Check-Up (FCU) (Experimental): Families recruited in Year 1 who are randomized to the FCU group will be provided with the Family Check-Up (FCU) after the initial in-home assessment and after 1 year follow-up assessment. The FCU is a brief (i.e., typically 3-5 sessions per year) family-centered intervention. The FCU intervention process consists of 3, and in some cases, 4 components: a) family assessment, b) a "Get to Know You" session, c) feedback, and d) follow-up treatment sessions.
  Interventions: Behavioral: Family Check-Up
- Waitlist Group (Experimental): Families recruited in Year 1 who are randomized to the wait-list group, and all families recruited in Year 2 will be assigned to the wait-list group. This group will receive the materials provided to all families, noted above, and the initial in-home assessment within 2 weeks of the screening to be conducted by a trained research assistant. At 1 year post-screening, the families in the wait-list group will be administered the follow-up assessment and will begin the Family Check-Up (FCU) intervention.
  Interventions: Behavioral: Family Check-Up
- Control Group (No Intervention): These families will be recruited in Year 3 of the study. These families will be provided the materials noted above and will receive the in-home assessments conducted by a trained research assistant. The initial in-home assessments will be conducted within 2 weeks of the screening, and follow-up assessments conducted 1 year post-screening.

INTERVENTIONS:
Behavioral: Family Check-Up — The Family Check-Up (FCU) is a brief, family-based program to prevent Substance Use/Substance Use Disorder (SU/SUD) with replicated efficacy
  Arms: Family Check-Up (FCU); Waitlist Group

SUMMARY:
This study is to test the effectiveness of integrating and adapting two National Institute on Drug Abuse (NIDA)-funded procedures for use in primary care pediatric clinics serving low-income youth: 1)the Youth Risk Index (YRI) and Transmissible Liability Index-Parent (TLI-P) nurse and/or research assistant-administered screening tools for high risk of substance use (SU) prior to high school and thus also for SUD and 2) the Family Check-Up (FCU) - a brief, family-based program to prevent SU/SUD with replicated efficacy.

DETAILED DESCRIPTION:
This study is to test the effectiveness of integrating and adapting two National Institute on Drug Abuse (NIDA)-funded procedures for use in primary care pediatric clinics serving low-income youth: 1) the Youth Risk Index (YRI) and Transmissible Liability Index (TLI-P) nurse and/or research assistant-administered screening tools for high risk of substance use (SU) prior to high school and thus also for SUD and 2) the Family Check-Up (FCU) - a brief, family-based program to prevent SU/SUD with replicated efficacy.

The following three aims focus on evaluating and refining the adaptation of the YRI & TLI-P program for primary-care use: 1) to replicate the effectiveness of the YRI & TLI-P screening tool in terms of concurrent and predictive validity and the engagement rate in the FCU; 2) to identify and address challenges in implementing and integrating the YRI & TLI-P/FCU prevention strategy within a primary care clinic serving urban, low-income youth; and 3) to test the effectiveness of the YRI & TLI-P/FCU on emerging SU, sexual activity, and conduct problems, as well as the putative mediators of these outcomes including parenting and parental well-being.

Based on prior FCU efficacy studies, 500 dyads of parents and their 9 years, 9 months to 13 years, 11 months old children from low-income, ethnically diverse families will be recruited from two large primary care clinics in an urban community. The FCU will be delivered for two or three years to test impact of dosage. Participants will be followed-up one year after completing FCU to evaluate longitudinal outcomes of the Integrated YRI & TLI-P/FCU .

ELIGIBILITY:
Inclusion Criteria:

* Child Aged 9 years, 9 months to 13 years, 11 months.
* A biological or adoptive parents or legal guardian with appropriate documentation with custody of the child.
* Either child or parent's score on screening assessment score must fall in elevated risk range.
* Child must be recipient of needs based Medicaid or family income must be at or below 150% Health and Human Services (HHS) Poverty Guidelines.

Exclusion Criteria:

* Inability to read English,
* Having moderate to severe mental disability (based on medical records),
* Child not accompanied by a biological or adoptive parent with legal custody or legal guardian with appropriate documentation
* Participant in the Early Steps Project

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 722 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Assessment of Liability and EXposure to Substance use and Antisocial behavior (ALEXSA) | baseline
  Administer Assessment of Liability and EXposure to Substance use and Antisocial behavior (ALEXSA)
Assessment of Liability and EXposure to Substance use and Antisocial behavior (ALEXSA) | twelve months
  Administer Assessment of Liability and EXposure to Substance use and Antisocial behavior (ALEXSA)
Assessment of Liability and EXposure to Substance use and Antisocial behavior (ALEXSA) | twenty-four months
  Administer Assessment of Liability and EXposure to Substance use and Antisocial behavior (ALEXSA)
Contextual Risk and Resources - 1 | baseline
  Administer Centers for Epidemiological Studies Depression Scale (CESD)
Contextual Risk and Resources - 1 | twelve months
  Administer Centers for Epidemiological Studies Depression Scale (CESD)
Contextual Risk and Resources - 1 | twenty-four months
  Administer Centers for Epidemiological Studies Depression Scale (CESD)
Contextual Risk and Resources - 2 | baseline
  Administer Demographic Questionnaire (DEMO)
Contextual Risk and Resources - 2 | twelve months
  Administer Demographic Questionnaire (DEMO)
Contextual Risk and Resources - 2 | twenty-four months
  Administer Demographic Questionnaire (DEMO)
Contextual Risk and Resources - 3 | baseline
  Administer Dyadic Adjustment Scale (DYAD)
Contextual Risk and Resources - 3 | twelve months
  Administer Dyadic Adjustment Scale (DYAD)
Contextual Risk and Resources - 3 | twenty-four months
  Administer Dyadic Adjustment Scale (DYAD)
Contextual Risk and Resources - 4 | baseline
  Administer Financial Stress Questionnaire (FINCE)
Contextual Risk and Resources - 4 | twelve months
  Administer Financial Stress Questionnaire (FINCE)
Contextual Risk and Resources - 4 | twenty-four months
  Administer Financial Stress Questionnaire (FINCE)
Contextual Risk and Resources - 5 | baseline
  Administer Me and My Neighborhood Questionnaire (MMNQ)
Contextual Risk and Resources - 5 | twelve months
  Administer Me and My Neighborhood Questionnaire (MMNQ)
Contextual Risk and Resources - 5 | twenty-four months
  Administer Me and My Neighborhood Questionnaire (MMNQ)
Contextual Risk and Resources - 6 | baseline
  Administer Parent Substance Use Questionnaire (SUBST-PC)
Contextual Risk and Resources - 6 | twelve months
  Administer Parent Substance Use Questionnaire (SUBST-PC)
Contextual Risk and Resources - 6 | twenty-four months
  Administer Parent Substance Use Questionnaire (SUBST-PC)
Youth Outcomes - 1 | baseline
  Administer Child Behavior Checklist (CBCL)
Youth Outcomes - 1 | twelve months
  Administer Child Behavior Checklist (CBCL)
Youth Outcomes - 1 | twenty-four months
  Administer Child Behavior Checklist (CBCL)
Youth Outcomes - 2 | baseline
  Assess Extracurricular Activities (ECA)
Youth Outcomes - 2 | twelve months
  Assess Extracurricular Activities (ECA)
Youth Outcomes - 2 | twenty-four months
  Assess Extracurricular Activities (ECA)
Youth Outcomes - 3 | baseline
  Administer Recent Activities Interview (RAI)
Youth Outcomes - 3 | twelve months
  Administer Recent Activities Interview (RAI)
Youth Outcomes - 3 | twenty-four months
  Administer Recent Activities Interview (RAI)
Youth Outcomes - 4 | baseline
  Administer Screen for Child Anxiety-Related Emotional Disorders (SCR)
Youth Outcomes - 4 | twelve months
  Administer Screen for Child Anxiety-Related Emotional Disorders (SCR)
Youth Outcomes - 4 | twenty-four months
  Administer Screen for Child Anxiety-Related Emotional Disorders (SCR)
Youth Outcomes - 5 | baseline
  Administer Self-Report of Delinquency (SHORT) (SRD)
Youth Outcomes - 5 | twelve months
  Administer Self-Report of Delinquency (SHORT) (SRD)
Youth Outcomes - 5 | twenty-four months
  Administer Self-Report of Delinquency (SHORT) (SRD)
Youth Outcomes - 6 | baseline
  Target Child Substance Use (TC Subst)
Youth Outcomes - 6 | twelve months
  Target Child Substance Use (TC Subst)
Youth Outcomes - 6 | twenty-four months
  Target Child Substance Use (TC Subst)
Youth Outcomes - 7 | baseline
  Administer Youth Risk Behavior Survey (YRBS)
Youth Outcomes - 7 | twelve months
  Administer Youth Risk Behavior Survey (YRBS)
Youth Outcomes - 7 | twenty-four months
  Administer Youth Risk Behavior Survey (YRBS)
Parenting and Family Socialization - 1 | baseline
  Evaluate using Adult Child Relationship scale (ACRS)
Parenting and Family Socialization - 1 | twelve months
  Evaluate using Adult Child Relationship scale (ACRS)
Parenting and Family Socialization - 1 | twenty-four months
  Evaluate using Adult Child Relationship scale (ACRS)
Parenting and Family Socialization - 2 | baseline
  Distressing Experiences Microaggression Scale (MIC)
Parenting and Family Socialization - 2 | twelve months
  Distressing Experiences Microaggression Scale (MIC)
Parenting and Family Socialization - 2 | twenty-four months
  Distressing Experiences Microaggression Scale (MIC)
Parenting and Family Socialization - 3 | baseline
  Child Daily Face-to-Face Racial Discrimination (CDIS)
Parenting and Family Socialization - 3 | twelve months
  Child Daily Face-to-Face Racial Discrimination (CDIS)
Parenting and Family Socialization - 3 | twenty-four months
  Child Daily Face-to-Face Racial Discrimination (CDIS)
Parenting and Family Socialization - 4 | baseline
  Assess using Parental Involvement Scale (PI)
Parenting and Family Socialization - 4 | twelve months
  Assess using Parental Involvement Scale (PI)
Parenting and Family Socialization - 4 | twenty-four months
  Assess using Parental Involvement Scale (PI)
Parenting and Family Socialization - 5 | baseline
  Parental Monitoring Interview - Parent Response, - Child Response (PMI-PR, PMI-CR)
Parenting and Family Socialization - 5 | twelve months
  Parental Monitoring Interview - Parent Response, - Child Response (PMI-PR, PMI-CR)
Parenting and Family Socialization - 5 | twenty-four months
  Parental Monitoring Interview - Parent Response, - Child Response (PMI-PR, PMI-CR)
Parenting and Family Socialization - 6 | baseline
  Assess using Parenting Children and Adolescents measure (PARCA)
Parenting and Family Socialization - 6 | twelve months
  Assess using Parenting Children and Adolescents measure (PARCA)
Parenting and Family Socialization - 6 | twenty-four months
  Assess using Parenting Children and Adolescents measure (PARCA)
Parenting and Family Socialization - 7 | baseline
  Assessment using Parental Rating of Peers and Social Skills (PPRSK)
Parenting and Family Socialization - 7 | twelve months
  Assessment using Parental Rating of Peers and Social Skills (PPRSK)
Parenting and Family Socialization - 7 | twenty-four months
  Assessment using Parental Rating of Peers and Social Skills (PPRSK)
Parenting and Family Socialization - Discussion Tasks - 1 | baseline
  Assessment using Parent Child Hot topics Discussion Task
Parenting and Family Socialization - Discussion Tasks - 1 | twelve months
  Assessment using Parent Child Hot topics Discussion Task
Parenting and Family Socialization - Discussion Tasks - 1 | twenty-four months
  Assessment using Parent Child Hot topics Discussion Task
Parenting and Family Socialization - Discussion Tasks - 2 | baseline
  Assessment using Parent Child Hot Topics Questionnaire (PCHT)
Parenting and Family Socialization - Discussion Tasks - 2 | twelve months
  Assessment using Parent Child Hot Topics Questionnaire (PCHT)
Parenting and Family Socialization - Discussion Tasks - 2 | twenty-four months
  Assessment using Parent Child Hot Topics Questionnaire (PCHT)
Parenting and Family Socialization - Discussion Tasks - 3 | baseline
  Assessment using Monitoring & Listening Discussion Task
Parenting and Family Socialization - Discussion Tasks - 3 | twelve months
  Assessment using Monitoring & Listening Discussion Task
Parenting and Family Socialization - Discussion Tasks - 3 | twenty-four months
  Assessment using Monitoring & Listening Discussion Task
Parenting and Family Socialization - Discussion Tasks - 4 | baseline
  Assessment using Recognition Discussion Task
Parenting and Family Socialization - Discussion Tasks - 4 | twelve months
  Assessment using Recognition Discussion Task
Parenting and Family Socialization - Discussion Tasks - 4 | twenty-four months
  Assessment using Recognition Discussion Task
Parenting and Family Socialization - Discussion Tasks - 5 | baseline
  Assessment using Family Culture Discussion Task

CONTACTS AND LOCATIONS:
Overall Officials: Ty Ridenour, PhD, Principal Investigator — RTI International
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galan CA, Meza JI, Ridenour TA, Shaw DS. Racial Discrimination Experienced by Black Parents: Enduring Mental Health Consequences for Adolescent Youth. J Am Acad Child Adolesc Psychiatry. 2022 Oct;61(10):1251-1261. doi: 10.1016/j.jaac.2022.04.015. Epub 2022 May 2. PMID 35513191